CLINICAL TRIAL: NCT00883532
Title: Prevention of Chronic Lung Disease (CLD) in Preterm Infants -A New Therapeutic Regimen
Brief Title: Prevention of Chronic Lung Disease (CLD) in Preterm Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Medical University Hospital (Other); Cathay General Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Tsu F. Yeh/ Chair professor of Pediatrics, College of medicine, china medical university,Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Yeh 2009 (CMU); NHRI
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2009-04

CONDITIONS: Respiratory Distress Syndrome; Chronic Lung Disease of Prematurity
Keywords: Preterm infant; Respiratory distress syndrome; chronic lung disease; budesonide; surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia; Premature Birth | interventions — Budesonide; Surface-Active Agents; Air; beractant

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- budesonide (Experimental): The treatment group will receive surfactant and budesonide.
  Interventions: Drug: budesonide
- surfactant and air (Placebo Comparator): The placebo group will receive surfactant and air as control.
  Interventions: Drug: surfactant and air (placebo)

INTERVENTIONS:
Drug: budesonide — budesonide, 0.25 mg/Kg/dose every 8 hours until the infant requires FIO2 < 30% or is extubated
  Other Names: pulmicort
  Arms: budesonide
Drug: surfactant and air (placebo) — receive surfactant and air as control through endotracheal route
  Other Names: survanta
  Arms: surfactant and air

SUMMARY:
Pulmonary inflammation plays an important role in the early development of CLD. Postnatal glucocorticoids have been shown effective in the prevention or treatment of CLD with various success. However, systemic glucocorticoid therapy often associated with various short term and long term complications. Therefore, modification of the therapeutic regimen is needed. Inhaled steroid, including inhaled budesonide,have been tried but the results are essentially unsuccessful, most likely due to small airways that the inhaled steroid reaching to the peripheral lungs are limited and unpredictable. Direct instillation of budesonide into the airway has also shown to be ineffective, possibly due to poor distribution of steroid in the lungs.

The investigators hypothesize that intratracheal instillation of budesonide, a strong tropical steroid, using surfactant as vehicle would facilitate the delivery of budesonide to the lung periphery and would inhibit lung inflammation and improve the pulmonary outcome. The result of our pilot study (Pediatrics, 2008) indicated this high possibility.

DETAILED DESCRIPTION:
After informed consent is obtained, infant will be randomly assigned to two groups based on a double-blind design. Group I will receive surfactant and budesonide and GII will receive surfactant and air as control through endotracheal route. Therapy will be given every 8 hours until the infant require FIO2 < 30% or is extubated. The end point of assessment is the combined incidence of CLD and death judged at 36 weeks postconceptional age and the long term neurological and cognitive function at 2-3 years.

The incidence of CLD and death in the selective group of infant is about 60%. Using this 60% incidence in the placebo group and expected 40% (33% improvement) in the treated group, 130 infants in each group is needed to detected a difference, permitting a 5% chance of type I error and 10% chance of type II error. The total safe target number will be 300; 150 in each group. A collaborative study is therefore proposed. The primary outcome to be assessed is the combined incidence of CLD and death. The secondary outcome to be assessed is short term and long term side effects.

ELIGIBILITY:
Inclusion Criteria:

* Infant with birth weight between 500-1500 gram
* Severe respiratory distress syndrome and requires mechanical ventilation with FIO2 > 60% shortly after birth

Exclusion Criteria:

* Severe congenital anomalities
* Lethal cardiopulmonary status at birth

Ages: 30 Minutes to 4 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Chronic lung disease morbidity among the survival | 36 postconceptional weeks

SECONDARY OUTCOMES:
Neurodevelopment | 2 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Tsu F Yeh, M.D., Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan, China

REFERENCES:
- [Background] Yeh TF, Lin HC, Chang CH, Wu TS, Su BH, Li TC, Pyati S, Tsai CH. Early intratracheal instillation of budesonide using surfactant as a vehicle to prevent chronic lung disease in preterm infants: a pilot study. Pediatrics. 2008 May;121(5):e1310-8. doi: 10.1542/peds.2007-1973. Epub 2008 Apr 21. PMID 18426851
- [Derived] Yeh TF, Chen CM, Wu SY, Husan Z, Li TC, Hsieh WS, Tsai CH, Lin HC. Intratracheal Administration of Budesonide/Surfactant to Prevent Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2016 Jan 1;193(1):86-95. doi: 10.1164/rccm.201505-0861OC. PMID 26351971
- See also: click here for more information about the study; prevention of chronic lung disease in preterm infants--a new therapeutic regimen — http://www.cmu.edu.tw